CLINICAL TRIAL: NCT05184595
Title: Cost-Utility Analysis of Home-based Versus Hospital-based Chemotherapy in Multiple Myeloma: Case of Carfilzomib
Acronym: ADHOMY2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pierre FEUGIER, Professor, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A00605-34
Record Dates: First submitted 2021-11-12; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Carfilzomib; Hospital-at-Home (HaH); Outpatient-Hospital (OH); Cost-Utility
MeSH Terms: conditions — Multiple Myeloma | interventions — hydroxide ion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carfilzomib delivered in OH only (Active Comparator): Patients receive the whole treatment in OH. Primary and secondary endpoints are collected at day 1 of cycle 3, 6, 9, 12, 18 and one month after.
  Patients leave the protocol prematurely due to treatment failure, toxicity or patient wishes. For those patients, the end of study visit will be done one month after ending treatment.
  Interventions: Other: Carfilzomib delivered in OH only
- Carfilzomib delivered in OH and HaH combined (Experimental): Patients receive the first cycle of treatment in OH. Then, they are randomized between exclusive OH treatment and combined treatment in OH and at home with HaH services.
  For the HaH patients group, the first injection of each cycle is delivered in OH. The rest of the cycle is delivered at home by HaH after a clinical examination (by nurse or general practitionner).
  Primary and secondary endpoints are collected at day 1 of cycle 3, 6, 9, 12, 18 and one month after.
  Patients leave the protocol prematurely due to treatment failure, toxicity or patient wishes. For those patients, the end of study visit will be done one month after ending treatment.
  Interventions: Other: Carfilzomib delivered in OH and HaH combined

INTERVENTIONS:
Other: Carfilzomib delivered in OH only — Patients receive the whole treatment en OH.
  Arms: Carfilzomib delivered in OH only
Other: Carfilzomib delivered in OH and HaH combined — Patients receive the first cycle of treatment in OH. Then, they are randomized between exclusive OH treatment and combined treatment in OH and at home with HaH services.
  Arms: Carfilzomib delivered in OH and HaH combined

SUMMARY:
Carfilzomib is administered in treatment of Multiple Myeloma intravenously on two consecutive days, each week for three weeks (days 1, 2, 8, 9, 15, and 16), followed by a 12-day rest period (days 17 to 28). With COVID pandemic, the investigators had to limit patient visits to the hospital. The treatment protocols were modified by switching to weekly injections of carfilzomib according to the PLEIADES and ARROW 2 studies.

Considering the frequency of intravenous (IV) administration, home-based chemotherapy in Hospital-at-Home (HaH) setting is an attractive and suitable alternative to standard hospital-based chemotherapy in Outpatient-Hospital (OH), and is expected to provide both cost-savings for the Health Insurance (HI) and improvement in patient quality of life (QoL).

The purpose of the study is to assess the cost-utility of home-based compared to hospital-based carfilzomib administration in multiple myeloma.

The investigators are also planning on assessing healthcare resource utilization and related costs, adverse and intercurrent events, and patients' quality of life and satisfaction, for each strategy.

DETAILED DESCRIPTION:
All participants receive the first cycle of treatment in OH. They are then randomized between exclusive OH treatment and combined treatment in OH and at home with HaH services.

For the HaH group, the first injection of each cycle is delivered in OH. The rest of the cycle is delivered at home by HaH after a clinical examination (by nurse or general practitionner).

Primary and secondary endpoints are collected at day 1 of cycle 3, 6, 9, 12, 18 and one month after the end of treatment.

Participants we leave the protocol prematurely in case of treatment failure, toxicity or if participant ask to. For those patients, the end of study visit will be done one month after ending treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* relapsed multiple myeloma, at least one prior line of treatment
* treatment with carfilzomib validated in a multidisciplinary consultation meeting and accepted by the patient
* The patient accepts mixed management and benefits from the support of his/her family and friends (see ANAES 2003 criteria). If the patient does not have a caregiver, he/she can still participate in the research and the absence of a caregiver will be collected.
* Patient capable of adhering to care (cf. ANAES 2003 criteria)
* Patient affiliated to a social security system or beneficiary of such a system.
* Patient having received full information on the organization of the research and having signed his or her informed consent

Exclusion Criteria:

* Person with a contraindication to carfilzomib
* Women of childbearing age who do not have effective contraception
* Persons referred to in articles L. 1121-5, L. 1121-7; L1121-8 and L1122-1-2 of the Public Health Code
* Pregnant woman, parturient or nursing mother
* Minor (not emancipated)
* Adult person under a legal protection measure (guardianship, curatorship, safeguard of justice)
* A person of full age who is unable to express his or her consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Incremental cost-utility ratio (ICUR) expressed in euros per QALY. | Up to 20 months
  Incremental cost-utility ratio (ICUR) of home-based compared to hospital-based carfilzomib administration in multiple myeloma, expressed in euros per QALY according to EQ-5D-5L questionnaire (EuroQOL 5 dimensions 5 levels) from 0 to 1 (1 being the best state with no problem)
Differences of quality of life in cancer patients between each group | Up to 20 months
  Difference of quality of life according to EORTC QLQ-C30 questionnaire (European Organisation for Research and Treatment of Cancer Quality of life Questionnaire with 30 questions, answer from 1 to 4, 1 being the best state with no problem)
Differences of quality of life in myeloma patients between each group | Up to 20 months
  Difference of quality of life according to EORTC QLQ-MY20 questionnaire (European Organisation for Research and Treatment of Cancer Quality of life Questionnaire with 20 questions related to myeloma symptoms, answer from 1 to 4, 1 being the best state with no problem)
Cost of care | Up to 20 month
  Cost for Health Insurance by patients, at the end of treament: Total costs per patient and average cost per injection

SECONDARY OUTCOMES:
Healthcare resource utilization | Up to 20 months
  * Rate of emergency visits to the Emergency Room
  * Rate of emergency consultation with the attending physician
  * Call rate in the referring center (Nancy Hospital)
Adverse events related to myeloma treatment | Up to 20 months
  * Rate of nosocomial infection, neuropathy, digestive disorders
  * Unscheduled hospitalization rates
Patients and caregivers' satisfaction | Up to 20 months
  - Patients' and Caregivers' Satisfaction Scores at the end of the treatment according to questionnaires with (opened and closes-questions) : 4 questions for OH group 9 questions for OH and HaH group 7 questions for caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FEUGIER, Principal Investigator — Central Hospital, Nancy, France